CLINICAL TRIAL: NCT05084859
Title: A Phase 1b, Open-Label, Dose-Escalation, Dose-Expansion Study Evaluating the Safety, Pharmacokinetics, and Efficacy of Orally Administered SM08502 Combined With Hormonal Therapy or Chemotherapy in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Preliminary Efficacy of Orally Administered SM08502 Combined With Hormonal Therapy or Chemotherapy in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due business reasons by Sponsor.
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SM08502-ONC-03
Record Dates: First submitted 2021-09-24; First posted 2021-10-20 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Castration-resistant Prostate Cancer; Non-small Cell Lung Cancer; Colorectal Cancer
Keywords: SM08502; pan Clk/Dyrk inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — abiraterone; Prednisone; Docetaxel; IFL protocol; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CRPC (Castration Resistant Prostate Cancer) - SM08502 + Abiraterone/Prednisone (Experimental): Part 1 (dose escalation cohorts) will evaluate SM08502 in subjects with advanced CRPC.
  Subjects will receive increasing doses of SM08502 with fixed doses of Abiraterone/Prednisone to determine the MTD and recommended Part 2 dose and schedule.
  Escalation will follow a 3+3+3 design within each cohort.
  Part 2 will further evaluate the recommended dose and schedule of SM08502 in subjects with advanced CRPC. Approximately 20 subjects will be enrolled.
  Interventions: Drug: SM08502; Drug: Abiraterone; Drug: Prednisone
- NSCLC (Non-Small Cell Lung Cancer) - SM08502 + Docetaxel (Experimental): Part 1 (dose escalation cohorts) will evaluate SM08502 in subjects with advanced NSCLC.
  Subjects will receive increasing doses of SM08502 with fixed doses of docetaxel to determine the MTD and recommended Part 2 dose and schedule.
  Escalation will follow a 3+3+3 design within each cohort.
  Part 2 will further evaluate the recommended dose and schedule of SM0850 in subjects with advanced NSCLC. Approximately 20 subjects will be enrolled.
  Interventions: Drug: SM08502; Drug: Docetaxel
- CRC (Colorectal Cancer) - SM08502 + FOLFIRI/Panitumumab (Experimental): Part 1 (dose escalation cohorts) will evaluate SM08502 in subjects with advanced CRC.
  Subjects will receive increasing doses of SM08502 with fixed doses of FOLFIRI plus panitumumab ( RAS wild type tumors) or with fixed doses of FOLFIRI (RAS mutant tumors)
  Escalation will follow a 3+3+3 design within each cohort.
  Part 2 will further evaluate the recommended dose and schedule of SM08502. Subjects that have RAS wild type tumors will receive FOLFIRI and panitumumab with SM08502 (n=15). Subjects that have RAS mutant tumors will receive FOLFIRI with SM08502 (n=15).
  Interventions: Drug: SM08502; Drug: FOLFIRI Protocol; Drug: Panitumumab

INTERVENTIONS:
Drug: SM08502 — SM08502 to be administered orally.
Drug: Abiraterone — Abiraterone to be administered orally.
  Arms: CRPC (Castration Resistant Prostate Cancer) - SM08502 + Abiraterone/Prednisone
Drug: Prednisone — Prednisone to be administered orally.
  Arms: CRPC (Castration Resistant Prostate Cancer) - SM08502 + Abiraterone/Prednisone
Drug: Docetaxel — Docetaxel to be administered intravenously.
  Arms: NSCLC (Non-Small Cell Lung Cancer) - SM08502 + Docetaxel
Drug: FOLFIRI Protocol — FOLFIRI Protocol to be administered intravenously.
  Arms: CRC (Colorectal Cancer) - SM08502 + FOLFIRI/Panitumumab
Drug: Panitumumab — Panitumumab to be administered intravenously.
  Arms: CRC (Colorectal Cancer) - SM08502 + FOLFIRI/Panitumumab

SUMMARY:
This study is an open-label, multi-center, dose-escalation, dose expansion study in adult subjects with advanced solid tumors. The study will evaluate the safety, tolerability, PK, and preliminary anti-tumor efficacy of SM08502 administered orally (PO), once daily (QD), following a 5 days on 2 days off treatment schedule in combination with chemotherapy or hormonal therapy. Alternative dosing schedules may be explored in Part 1 if necessary. The recommended Part 2 dose and schedule for each combination will then be further evaluated in the Part 2 expansion.

Dosing will occur in 21- or 28-day cycles (depending on the combination partner) and treatment with SM08502 will continue within each subject unless treatment is discontinued due to toxicity, disease progression, initiation of a new anti-neoplastic therapy, withdrawal of consent, the Sponsor terminates the study, or the subject no longer meets retreatment criteria.

ELIGIBILITY:
Key Inclusion Criteria:

1.0. Part 1 - Subjects with advanced and/or metastatic solid tumors. Histologic or cytologic confirmation of malignancy must have been obtained at diagnosis. The tumor types include:

i. CRPC - Subjects with progressive disease in the setting of medical or surgical castration (i.e., castration-resistant prostate cancer).

ii. NSCLC (adenocarcinoma subtype) - Subjects with no targetable mutations must have received a platinum-containing doublet chemotherapy regimen and a checkpoint inhibitor (either in combination or monotherapy, if indicated) and have progressed. Subjects with targetable mutations/alterations such as EGFR, ALK, or NTRK must have received prior targeted therapy and have progressed.

iii. CRC - Subjects must have received one prior line of standard chemotherapy such as FOLFOX +/- a VEGF-inhibitor and have progressed or are intolerant of oxaliplatin based regimens.

1.1. Part 2 - Subjects with advanced and/or metastatic solid tumors. Histologic or cytologic confirmation of malignancy must have been obtained at diagnosis. The tumor types include:

i. CRPC - Subjects with progressive disease in the setting of medical or surgical castration (i.e., castration- resistant prostate cancer). Subjects who have not received chemotherapy, are not candidates for chemotherapy, or refuse chemotherapy are eligible (Arm A). Subjects who have received chemotherapy are eligible (Arm B), however, more than 2 prior lines of chemotherapy in any setting are excluded.

ii. NSCLC (adenocarcinoma subtype) - Subjects with no targetable mutations must have received a platinum-containing doublet chemotherapy regimen and a checkpoint inhibitor (either in combination or monotherapy, if indicated) and have progressed. Subjects with targetable mutations/alterations such as EGFR, ALK, NTRK must have received prior targeted therapy and have progressed.

iii. CRC - Subjects must have received one prior line of standard chemotherapy such as FOLFOX +/- either a VEGF-inhibitor or EGFR inhibitor (if indicated) and have progressed or are intolerant of oxaliplatin based regimens.

2.0. Male or female subjects ≥ 18 years of age.

3.0 Measurable or evaluable disease per RECIST 1.1 (Part 1). For Part 2, at least one measurable lesion per RECIST 1.1 that has not been previously irradiated. In CRPC subjects (Parts 1 and 2) without measurable disease per RECIST 1.1, a PSA that is concordant with clinical disease progression (rising) is eligible. A PSA value of 2 ng/ml or greater is required for study entry for those without measurable disease.

4.0. Subjects must have archived tumor specimens available for analysis Otherwise, a fresh tumor biopsy will be required at study entry.

5.0.. Subjects must have recovered (i.e., Grade 1 [or better] based on CTCAE v5.0) from all toxicity associated with previous chemotherapy, targeted therapy, experimental therapy, biological therapy, immuno-oncology therapy, surgery, radiotherapy, or other locoregional therapy.

The following intervals must elapse between end of last treatment and receiving the first dose of SM08502:

* Chemotherapy: 3 weeks.
* Mitomycin C or a nitrosourea: 6 weeks.
* Radiotherapy: 3 weeks.
* Major surgery: 6 weeks.
* Targeted therapy, including monoclonal antibodies and immuno-oncology therapies: 4 weeks or 5 half-lives, whichever is shortest.

6.0. Subjects must meet the following laboratory criteria at Screening for study entry:

* Hepatic function: serum total bilirubin ≤ 1.5x upper limit of normal (ULN), AST/ALT ≤ 2.5x ULN. For subjects with Gilbert's syndrome, serum total bilirubin ≤ 3x ULN.
* Renal function: measured or calculated creatinine clearance via Cockcroft-Gault formula >35 mL/min.
* Hematology: absolute neutrophil counts ≥ 1500/mm3, platelet counts ≥ 100,000/mm3, hemoglobin ≥ 9.0 g/dL.
* Coagulation: prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5x ULN.

7.0. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.

8.0. Life expectancy > 3 months.

9.0. Subjects must have no uncontrolled intercurrent illness.

10.0 Subjects must have the ability to swallow and retain oral medication.

11.0 Subjects must be willing to sign and provide informed consent and be capable of giving informed consent in accordance with the Institutional Review Board (IRB) / Ethics Committee (EC) policy.

Key Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Women of childbearing potential (WOCBP) must agree to follow the contraceptive guidelines as outlined in protocol.
3. Men of reproductive potential must agree to follow the contraceptive guidelines as outlined in protocol.
4. Subjects with a QTc (Fridericia's) prolongation > CTCAE v5.0 Grade 1 (>480 msec) at Screening.
5. Subjects with clinically significant ventricular tachycardia (VT), atrial fibrillation (AF), ventricular fibrillation (VF), second- or third-degree heart block.
6. Subjects with myocardial infarction (MI) within 1 year, Class II-IV congestive heart failure (CHF) per New York Heart Association (NYHA) classification, or clinically significant coronary artery disease (CAD)..
7. Subjects with active infection (e.g., requiring antibiotic therapy).
8. Organ transplant recipients.
9. Subjects with untreated, progressing, or known symptomatic brain metastasis.
10. Subjects with a second malignancy unless adequately treated with no recurrence for 3 years. Subjects with a history of previous or recent adequately treated basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of any source are eligible.
11. Subjects with known hypersensitivity to any excipients in the study drug formulation.
12. Subjects with active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of SM08502 per Investigator's opinion.
13. Subjects with known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection.
14. Subjects considered by the Investigator to be unsuitable for the study for any other reason.
15. Subjects with chronic liver disease or dysfunction and a Child-Pugh score of B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Part 1 - Incidence of Treatment Emergent Adverse Events (TEAEs) | Consent date to 28 days after the last dose of study treatment
  As measured by NCI CTCAE version 5.0.
Part 1 - Maximum tolerated dose (MTD) of SM08502 when combined with standard of care agents. | DLT period of 21 or 28 days per dose level depending on cycle length
  Based on frequency and severity of dose-limiting toxicities (DLTs).
Part 1 - Blood samples for measurement of the plasma levels of SM08502 and its metabolite | Sample collection timepoints: Cycle1 (Day1 (0,2,4,6, hrs), Day2, Day8, Day15, Day22) Cycle 2 (Day1, Day2) Cycle3-5 (Day1) and EOT. Each cycle is 21 or 28 days depending on tumor type.
  Maximum (Cmax) and minimum (Cmin) Plasma concentration of SM08502 and its metabolite SM08955.
Part 1 - Blood samples for measurement of the plasma levels of SM08502 and its metabolite | Sample collection timepoints: Cycle1 (Day1 (0,2,4,6, hrs), Day2, Day8, Day15, Day22) Cycle 2 (Day1, Day2) Cycle3-5 (Day1) and EOT. Each cycle is 21 or 28 days depending on tumor type.
  Area under the plasma concentration time curve (AUC) from zero to 24 hours: AUC0-24 for SM08502 and its metabolite SM08955
Part 1 - Blood samples for measurement of the plasma levels of SM08502 and its metabolite | Sample collection timepoints: Cycle1 (Day1 (0,2,4,6, hrs), Day2, Day8, Day15, Day22) Cycle 2 (Day1, Day2) Cycle3-5 (Day1) and EOT. Each cycle is 21 or 28 days depending on tumor type.
  Area under the plasma concentration time curve (AUC) from zero to the last measurable concentration: AUClast for SM08502 and its metabolite SM08955.
Part 1 - Plasma drug concentration | Sample collection timepoints: Cycle1 (Day1 (0,2,4,6, hrs), Day2, Day8, Day15, Day22) Cycle 2 (Day1, Day2) Cycle3-5 (Day1) and EOT. Each cycle is 21 or 28 days depending on tumor type.
  Maximum steady-state plasma drug concentration (Cmaxss) during a dosage interval.
Part 2 - Incidence of Safety and tolerability of SM08502 | Consent date to 28 days after the last dose of study treatment
  As measured by treatment emergent adverse events (TEAEs) as measured by NCI CTCAE version 5 from subjects treated at the recommended Part 2 dose and schedule.
Part 2 - Objective response rate | Approximately 5 years
  Using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or Prostate Cancer Working Group 3 Criteria (PCWG3) where appropriate.

SECONDARY OUTCOMES:
Part 1 - Objective Response rate | Approximately 5 years
  Tumor response using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or Prostate Cancer Working Group 3 Criteria (PCWG3) where appropriate.
Part 2 - Blood samples for measurement of the plasma levels of SM08502 and its metabolite | Sample collection timepoints: Cycle1 (Day1 (0,2,4,6, hrs), Day2, Day8, Day15,) Cycle 2-5 (Day1). Each cycle is 21 or 28 days depending on tumor type.
  Maximum (Cmax) and minimum (Cmin) Plasma concentration of SM08502 and its metabolite SM08955.
Part 2 - Blood samples for measurement of the plasma levels of SM08502 and its metabolite | Sample collection timepoints: Cycle1 (Day1 (0,2,4,6, hrs), Day2, Day8, Day15,) Cycle 2-5 (Day1). Each cycle is 21 or 28 days depending on tumor type.
  Area under the plasma concentration time curve (AUC) from zero to 24 hours: AUC0-24 for SM08502 and its metabolite SM08955
Part 2 - Blood samples for measurement of the plasma levels of SM08502 and its metabolite | Sample collection timepoints: Cycle1 (Day1 (0,2,4,6, hrs), Day2, Day8, Day15,) Cycle 2-5 (Day1). Each cycle is 21 or 28 days depending on tumor type.
  Area under the plasma concentration time curve (AUC) from zero to the last measurable concentration: AUClast for SM08502 and its metabolite SM08955.
Part 2 - Blood samples for measurement of the plasma levels of SM08502 and its metabolite | Sample collection timepoints: Cycle1 (Day1 (0,2,4,6, hrs), Day2, Day8, Day15,) Cycle 2-5 (Day1). Each cycle is 21 or 28 days depending on tumor type.
  Maximum steady-state plasma drug concentration (Cmaxss) during a dosage interval.

CONTACTS AND LOCATIONS:
Overall Officials: Darrin Beaupre, MD, PhD, CMO, Study Chair — Biosplice Therapeutics, Inc.
Locations (20):
- United States (16):
  - The University of Arizona Cancer Center (UACC) - North Campus, Tucson, Arizona
  - University of Colorado, Anschutz, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Cancer Institute (DCI) - Duke Cancer Center, Durham, North Carolina
  - The Carl and Edyth Lindner Center for Research and Education at The Christ Hospital, LLC, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology-San Antonio Northeast, San Antonio, Texas
  - UT Health San Antonio - Mays Cancer Center - Institute for Drug Development, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Seattle Cancer Care Alliance (SCCA), Seattle, Washington
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown
  - Saint Vincent's Hospital, Darlinghurst
  - Icon Cancer Care-South Brisbane, South Brisbane
  - The Queen Elizabeth Hospital (TQEH), Woodville South

IPD SHARING:
Plan to Share IPD: No